CLINICAL TRIAL: NCT00579514
Title: Germline Alterations of Tumor Susceptibility Genes in New York Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other); Weill Medical College of Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00-014
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Bladder Cancer; Kidney Cancer; Colon Cancer; Prostate Cancer; Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Ovarian Neoplasms

ARMS (2):
- 1 (Active Comparator): All incident second primary cancers of colon, breast, bladder, kidney, prostate, ovarian cancer lung cancer and lymphoid cancer diagnosed between 1999 and present will be included in the secondary design to compare second primary cancer "cases" and first primary "controls".
  Interventions: Genetic: PCR/PCR/LDR Strategy
- 2 (Placebo Comparator): Controls will be volunteer blood donors from the New York Blood Center as well as normal volunteers from other AMDeC sites.
  Interventions: Genetic: PCR/PCR/LDR Strategy

INTERVENTIONS:
Genetic: PCR/PCR/LDR Strategy — Evaluate the extent to which polymorphisms in BRCA1, BRCA2, PTEN, T β R1, TGF β-1, DNA repair genes (including ATM and CHK2), APC, ER, PR, MCP-1, MPIF, CCR2/5 and CCR3 are correlated with cancer incidence. Candidate genes will also be selected from 1) cytokine signaling and 2) apoptosis regulatory pathways.

SUMMARY:
The basic premise of this research proposal is to determine whether there is any significant association between germline polymorphisms and cancers of colon, bladder, breast, testicular, prostate, ovaries, kidney, lung, lymphoid organs, and head and neck. This is an exploratory study designed to generate hypotheses for further research.

DETAILED DESCRIPTION:
To establish significant correlations between genetic polymorphisms and cancer, a largescale, systematic comparison of genetic alterations utilizing a case-control methodology is proposed. To date, such studies have been limited due to the large number of samples necessary for obtaining statistical significance, and the lack of rapid and accurate methods to screen for genetic polymorphisms. We propose to utilize an anonymized design to obtain DNA from residual material from routine diagnostic blood tests, to link these samples to a limited set of clinical variables, and to test for the frequency of candidate low-penetrance cancer susceptibility alleles. These data will be combined with similar data from a control group of age- and ethnically-matched volunteers for a related cohort study to be conducted separately. Polymorphisms to be screened for include those involving the genes PTEN, APC, TGF βR-I, BLM, CHK2, a p85 phosphoprotein, ATM, ER, PR, MCP-1, MPIF, CCR2/5, CCR3, and SULT1A1. Cancers to be included are breast, bladder, kidney,colon, testicular, lung, prostate, ovarian, lymphoid neoplasms, and head and neck carcinomas. Genes with SNPs known to be relevant for either the development or treatment of lymphoid malignancies will also be targeted. Specifically, candidate genes will be selected from 1) cytokine signaling, 2) DNA repair, and 3) apoptosis regulatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of cancer of the colon, breast, bladder, kidney, testicles, lungs, prostate, head and neck, or lymphoid organs, who have donated a diagnostic blood sample as either an inpatient or outpatient at MSKCC.
* All patients who have two or more histologic diagnoses of the same primary tumor type involving the above sites.
* Patients of Ashkenazi Jewish ancestry with a histologic diagnosis of cancer of any type.
* Samples ascertained as part of protocol 98-024A(1) are also eligible for ascertainment in this study.

Exclusion Criteria:

* MSKCC patients without a histologic diagnosis of cancer of the breast, bladder, kidney, colon, testicles, lungs, prostate, or lymphoid malignancy (including all types of lymphoma) will not be eligible for the AMDeC sponsored component of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21081 (Actual)
Dates: Start 2000-03; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To collect anonymized germline DNA from patients with breast, bladder, kidney, lung, colon, testicular, prostate, lymphoid, ovarian or head and neck cancers, as well as patients with multiple primary cancers, from select New York City ethnic groups. | 20 years

SECONDARY OUTCOMES:
To analyze DNA samples from matched non-cancer individuals of the same ethnic groups available as part of the AMDeC-sponsored New York Cancer Study. | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org